CLINICAL TRIAL: NCT06571279
Title: Assessing the Impact of a Plant-Based Diet for Diabetes Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jean L. Fry (Other)
Responsible Party: Sponsor-Investigator, Jean L. Fry, Assistant Professor- PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 95349
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Prediabetes (Insulin Resistance, Impaired Glucose Tolerance)
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Glucose Intolerance | interventions — Diet, Plant-Based

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plant-based diet (Other): 5 weeks of plant-based meals and snacks.
  Interventions: Other: Plant-based diet

INTERVENTIONS:
Other: Plant-based diet — Standard plant-based meals will be provided directly to participants. The dietary intervention will begin with a one-week Western diet run-in; hereafter, participants will consume plant-based meals for approximately 5 weeks. Total energy provided will be equal to REE X 1.4 to account for light physical activity to support weight maintenance. High-inositol snacks will be provided to meet energy needs. Meals and snacks combined will provide a minimum of 20mg total inositol/kg body weight. For example, a 200lb participant will consume 1.8g daily, which is consistent with doses used in prior studies.

SUMMARY:
The primary purpose of this study is to determine the sex-specific metabolic and molecular response, among adults with prediabetes, when moving from a Western Diet to plant-based diet.

DETAILED DESCRIPTION:
Plant-based diets that are abundant in myoinsitol and D-chiro inositol (MI and DCI) increase insulin sensitivity by promotion of insulin signaling lowering serum insulin and improving insulin resistance. The Western diet contributes to chronic metabolic inflammation often leading to the development of metabolic diseases. There is known metabolic improvement among men compared to women when following a plant-based diet or intensive lifestyle modifications. Through this study we look to identify the pathways in which plant-based diet impact skeletal muscle inositol metabolites among sexes (men vs. women) and improve insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index greater than or equal to 27
* High waist circumference (women greater than or equal to 35"; men greater than or equal to 40")
* Prediabetes (based on fasting glucose 100-125 mg/dL, HbA1c 5.7-6.4, or 2-hr post-oral glucose tolerance test glucose screen between 140-199mg/dL)
* Physical activity below national guidelines
* Aged 30-55 (premenopausal for women)
* Following a Western diet

Exclusion Criteria:

* Diabetes diagnosis
* Take medications that may affect insulin sensitivity
* More than 5% weight change within 6 months of screening
* History of bariatric surgery
* Report any dietary supplement, medication, or medical condition known to significantly affect weight or metabolism
* Take hormone replacement therapy
* Consume 3 or more servings of combined fruit and vegetables daily and/or 3 or more servings of whole grains daily
* Any food allergy more severe than grade 1 on the CoFAR Grading Scale for Systemic Allergic Reactions, Version 3.0 or allergy to lidocaine

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since sex hormones may play a role in diet response, prospective participants taking a medication that significantly affects sex hormones (like estrogen or testosterone) will not be eligible to participate.
Enrollment: 9 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity (glucose infusion rate) | The first measure is taken immediately after the run-in and the final measure will be taken immediately after the completion of the plant-based diet intervention five weeks later.
  This gold standard test for IS will be performed at baseline and post-intervention with support of the COBRE Phenotyping core. After ≥8 hour fast, participants will be admitted to our Center for Clinical and Translational Science (CCTS) and two IVs inserted; one for infusion, the other for blood draws (see Phenotyping core). The primary outcome is the glucose infusion rate (GIR), a direct measure of whole body IS, which will enable us to detect even small changes in IS in response to the intervention. COBRE mentor Dr. Kern is proficient in use of these methods The primary clinical outcome is the change in GIR from post run-in to post intervention.
Skeletal muscle d-chiroinositol content | The first measure is taken immediately after the run-in and the final measure will be taken immediately after the completion of the plant-based diet intervention five weeks later.
  Muscle samples will be homogenized, then inositol compounds will be extracted using solvents. In the prepared samples, D-chiroinositol content will be assessed by a commercial service using LC-MS/MS.

SECONDARY OUTCOMES:
Phosphorylation status of insulin signaling molecules in skeletal muscle | The first measure is taken immediately after the run-in and the final measure will be taken immediately after the completion of the plant-based diet intervention five weeks later.
  Upon insulin stimulation, insulin-responsive signaling proteins are phosphorylated to initiate downstream effects. The ratio of phosphorylated and unphosphorylated, as well as total protein, per standard unit of skeletal muscle will be determined.
Absolute change in visceral fat (g) | The first measure is taken immediately after the run-in and the final measure will be taken immediately after the completion of the plant-based diet intervention five weeks later.
  Computed tomography will be used to measure visceral fat
Fasting blood glucose | The first measure is taken immediately after the run-in and the final measure will be taken immediately after the completion of the plant-based diet intervention five weeks later.
  Baseline measure of fasting blood glucose are measured via YSI before the start of the OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Jean L Fry, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky CCTS, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bedard A, Riverin M, Dodin S, Corneau L, Lemieux S. Sex differences in the impact of the Mediterranean diet on cardiovascular risk profile. Br J Nutr. 2012 Oct 28;108(8):1428-34. doi: 10.1017/S0007114511006969. Epub 2012 Jan 6. PMID 22221517
- [Background] Chen Z, Zuurmond MG, van der Schaft N, Nano J, Wijnhoven HAH, Ikram MA, Franco OH, Voortman T. Plant versus animal based diets and insulin resistance, prediabetes and type 2 diabetes: the Rotterdam Study. Eur J Epidemiol. 2018 Sep;33(9):883-893. doi: 10.1007/s10654-018-0414-8. Epub 2018 Jun 8. PMID 29948369
- [Background] Perreault L, Ma Y, Dagogo-Jack S, Horton E, Marrero D, Crandall J, Barrett-Connor E; Diabetes Prevention Program. Sex differences in diabetes risk and the effect of intensive lifestyle modification in the Diabetes Prevention Program. Diabetes Care. 2008 Jul;31(7):1416-21. doi: 10.2337/dc07-2390. Epub 2008 Mar 20. PMID 18356403
- [Background] Leblanc V, Begin C, Hudon AM, Royer MM, Corneau L, Dodin S, Lemieux S. Gender differences in the long-term effects of a nutritional intervention program promoting the Mediterranean diet: changes in dietary intakes, eating behaviors, anthropometric and metabolic variables. Nutr J. 2014 Nov 22;13:107. doi: 10.1186/1475-2891-13-107. PMID 25416917
- [Background] Sargrad KR, Homko C, Mozzoli M, Boden G. Effect of high protein vs high carbohydrate intake on insulin sensitivity, body weight, hemoglobin A1c, and blood pressure in patients with type 2 diabetes mellitus. J Am Diet Assoc. 2005 Apr;105(4):573-80. doi: 10.1016/j.jada.2005.01.009. PMID 15800559
- [Background] Bedard A, Tchernof A, Lamarche B, Corneau L, Dodin S, Lemieux S. Effects of the traditional Mediterranean diet on adiponectin and leptin concentrations in men and premenopausal women: do sex differences exist? Eur J Clin Nutr. 2014 May;68(5):561-6. doi: 10.1038/ejcn.2014.27. Epub 2014 Mar 5. PMID 24595221
- [Background] Minambres I, Cuixart G, Goncalves A, Corcoy R. Effects of inositol on glucose homeostasis: Systematic review and meta-analysis of randomized controlled trials. Clin Nutr. 2019 Jun;38(3):1146-1152. doi: 10.1016/j.clnu.2018.06.957. Epub 2018 Jun 21. PMID 29980312
- [Background] Soldevila-Domenech N, Pastor A, Sala-Vila A, Lazaro I, Boronat A, Munoz D, Castaner O, Fagundo B, Corella D, Fernandez-Aranda F, Martinez-Gonzalez MA, Salas-Salvado J, Fito M, de la Torre R. Sex differences in endocannabinoids during 3 years of Mediterranean diet intervention: Association with insulin resistance and weight loss in a population with metabolic syndrome. Front Nutr. 2022 Dec 1;9:1076677. doi: 10.3389/fnut.2022.1076677. eCollection 2022. PMID 36532543
- [Background] Brennan L, Gibbons H. Sex matters: a focus on the impact of biological sex on metabolomic profiles and dietary interventions. Proc Nutr Soc. 2020 May;79(2):205-209. doi: 10.1017/S002966511900106X. Epub 2019 Jul 31. PMID 31362802
- [Background] Larner J, Brautigan DL, Thorner MO. D-chiro-inositol glycans in insulin signaling and insulin resistance. Mol Med. 2010 Nov-Dec;16(11-12):543-52. doi: 10.2119/molmed.2010.00107. Epub 2010 Aug 27. PMID 20811656